CLINICAL TRIAL: NCT00408681
Title: A Pilot Study to Evaluate the Potential Efficacy of Lithium Carbonate for Stimulation of Intestinal Recovery In Patients With Acute Graft-versus-host Disease (GVHD)
Brief Title: Lithium Carbonate in Treating Patients With Acute Intestinal Graft-Versus-Host-Disease (GVHD) After Donor Stem Cell Transplant
Acronym: GVHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Martin, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2080.00; NCI-2010-00269
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, Breakpoint Cluster Region-abl Translocation (BCR-ABL) Negative; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Disseminated Neuroblastoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Gastrointestinal Complications; Juvenile Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Poor Prognosis Metastatic Gestational Trophoblastic Tumor; Previously Treated Childhood Rhabdomyosarcoma; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Neuroblastoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Small Lymphocytic Lymphoma; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage II Ovarian Epithelial Cancer; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Malignant Testicular Germ Cell Tumor; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Ovarian Epithelial Cancer; Stage III Small Lymphocytic Lymphoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Breast Cancer; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Ovarian Epithelial Cancer; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Wilms Tumor; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms | interventions — Lithium Carbonate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive oral lithium carbonate once or twice daily. Treatment continues for up to 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lithium carbonate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lithium carbonate — Given orally
  Other Names: Eskalith; Lithane; Lithium; Lithobid; Lithonate; Lithotabs
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Lithium carbonate may be an effective treatment for intestinal graft-versus-host disease caused by a donor stem cell transplant.

PURPOSE: This clinical trial is studying lithium carbonate in treating patients with acute intestinal graft-versus-host-disease after donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effects of lithium on functional and mucosal anatomic recovery in the small or large bowel of patients with acute GVHD.

II. Functional recovery will be evaluated according to changes in clinical manifestations of gastrointestinal GVHD. III. Mucosal anatomic recovery will be evaluated by review of results from clinically indicated endoscopic evaluations.

SECONDARY OBJECTIVES:

I. To assess the tolerability of lithium administration in allogeneic hematopoietic cell transplant recipients.

OUTLINE: Patients receive oral lithium carbonate once or twice daily. Treatment continues for up to 8 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of severe intestinal GVHD that is not improving at any time after initial treatment with glucocorticoids for at least 7 days are eligible for enrollment; measures indicating severity of GVHD will include: a) persistent diarrhea with average daily stool volumes > 500 mL per day; or b) persistent hemorrhage that is detectable by visual inspection of the stool
* Patients with denuded mucosa caused by GVHD are eligible for enrollment, regardless of prior treatment for acute GVHD; denuded mucosa is defined as loss (i.e., erosion or sloughing) of the epithelium in: a) at least one-third of the surface area in a 30 cm colonic segment (i.e., rectosigmoid, descending or transverse colon); or b) at least one fifth of the surface area of the second portion of the duodenum, as estimated by endoscopic evaluation; denuded mucosa must be documented by images of the duodenum and colon and by histologic evaluation of the colon
* All subjects must provide written informed consent with the use of forms approved by the Fred Hutchinson Cancer Research Center (FHCRC) Institutional Review Board (IRB)

Exclusion Criteria:

* Significant renal dysfunction (estimated creatinine clearance < 30 mL/min)
* Persistent or recurrent malignancy
* Secondary malignancy
* Patients who had autologous or syngeneic marrow transplantation
* Presence of any cause of intestinal symptoms or ulceration other than GVHD
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol will be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2010-11 (Actual); Study Completion 2015-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Martin, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Steinbach G, Hockenbery DM, Huls G, Furlong T, Myerson D, Loeb KR, Fann JR, Castilla-Llorente C, McDonald GB, Martin PJ. Pilot study of lithium to restore intestinal barrier function in severe graft-versus-host disease. PLoS One. 2017 Aug 17;12(8):e0183284. doi: 10.1371/journal.pone.0183284. eCollection 2017. PMID 28817727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with severe gastrointestinal acute graft-versus-host disease with or without mucosal denudation identified by endoscopy were recruited from a hospitalized population of patients who had recent allogeneic hematopoietic cell transplantation.
Pre-assignment Details: Patients were enrolled according to eligibility criteria in the protocol.
Groups:
- Treated Patients: Patients receive oral lithium carbonate once or twice daily orally. Treatment continues for up to 8 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treated Patients
Started | 20
Completed | 11 (Completion was defined as administration of the study product for at least 28 days.)
Not Completed | 9
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Groups:
- Treated Patients: Patients received oral lithium carbonate once or twice daily. Treatment continued for up to 8 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [22 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 14
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Indication for transplantation [Count of Participants; unit: Participants]
  Non-Hodgkin lymphoma | 3
  Acute myeloid leukemia | 6
  Multiple myeloma | 2
  Chronic myeloid leukemia | 2
  Acute lymphoid leukemia | 3
  Myelodysplastic syndrome | 1
  Aplastic anemia | 1
  Paroxysmal nocturnal hemoglobinuria | 1
  Chronic lymphocytic leukemia | 1
Type of pretransplant conditioning regimen [Count of Participants; unit: Participants]
  Myeloablative | 12
  Nonmyeloablative | 8
Graft-versus-host disease (GVHD) prophylaxis regimen [Count of Participants; unit: Participants]
  Cyclosporine and mycophenolate mofetil (MMF) | 8
  Tacrolimus and methotrexate | 10
  Cyclophosphamide, tacrolimus, MMF | 1
  Tacrolimus and mycophenolate mofeftil | 1
Mucosal denudation [Count of Participants; unit: Participants]
  Duodenum alone | 7
  Colon alone | 7
  Duodenum and colon | 3
Agents given to prevent GVHD at the time of enrollment [Count of Participants; unit: Participants]
  Tacrolimus | 8
  Cyclosporine | 7
  Mycophenolate mofetil | 8
Agents given to treat GVHD more than 3 days before enrollment in the study [Count of Participants; unit: Participants]
  Infliximab | 3
  Rabbit anti-thymocyte globulin | 3
  Horse anti-thymocyte globulin | 1
  Extracorporeal photopheresis | 2
  Mesenchymal stem cells | 1
  Mycophenolate mofetil | 5
  Tacrolimus | 3
  Sirolimus | 1
  Cyclosporine | 1
Interval from transplantation to start of study product administration [Median (Full Range); unit: days] | 90 [22 to 215]
Agents given to treat GVHD within 3 days before or after enrollment [Count of Participants; unit: Participants]
  Methotrexate | 1
  Pentostatin | 2
  Rabbit anti-thymocyte globulin | 4
  Mycophenolate mofetil | 1
  Infliximab | 2
  Alemtuzumab | 1

OUTCOME MEASURES:

1. Primary Outcome: Functional Recovery
Description: Functional recovery was defined as partial or complete resolution of gastrointestinal manifestations of acute graft-versus-host disease. Gastrointestinal manifestations of acute graft-versus-host disease include anorexia, nausea, vomiting, diarrhea, abdominal pain and bleeding. Complete response (CR) of intestinal GVHD was defined as the absence of any symptoms referable to intestinal GVHD. Partial response (PR) was defined as clearing of abdominal pain (or withdrawal of opioid analgesic requirements in patients treated for abdominal pain) and of grossly visible bleeding if present, and resolution of diarrhea or decrease in the three day average stool volume by ≥ 500 mL in patients with stool volumes of ≥ 500 mL. Progression of GVHD was defined as an increase in the three day average stool volume by > 500 mL, or the development of new abdominal pain (or new opioid analgesic requirements) or new intestinal bleeding.
Time Frame: at 28 days after starting treatment with the study product
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants
  Complete clinical response | 10
  Partial clinical response | 1
  No response or clinical progression | 6
  Death before day 28 | 3

2. Secondary Outcome: Duration of Treatment With the Study Product
Description: Number of days from beginning of orally administered lithium carbonate to the end of orally administered lithium carbonate
Time Frame: Up to 6 months
Measure: Median (Full Range); unit: days
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
days | 30.5 [7 to 172]

3. Secondary Outcome: Mucosal Anatomic Recovery
Description: Endoscopic evaluation of improvement. Categories include 1) no improvement, 2) regenerative changes, 3) limited improvement, 4) partial improvement and 5) complete response. Endoscopic manifestations of acute graft-versus-host disease include edema, erythema, mucosal ulceration and denudation. Complete mucosal recovery was defined as the appearance of intact mucosa with at least 98% of the luminal surface covered by epithelium. Partial response was defined as the appearance of mostly intact mucosa with at least 80% improvement or less than 10% denuded. Limited response was retrospectively designated to describe visible improvement that was less than partial response. Regenerative change was retrospectively designated to describe early reappearance of mucosal integrity in a previously denuded area but not sufficient to meet criteria for partial response. Failure to respond was defined as failure to meet partial response criteria.
Time Frame: 2 to 3 weeks after starting treatment with the study product
Population: Only 8 of the 20 enrolled patients had endoscopic evaluation during this time window.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 8
Participants
  No improvement | 3
  Regenerative changes | 3
  Partial improvement | 2

4. Secondary Outcome: Mucosal Anatomic Recovery
Description: as for outcome 3
Time Frame: 4 weeks after starting treatment with the study product
Population: Only 2 patients had endoscopic evaluation during this time window.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 2
Participants
  Limited improvement | 1
  Partial improvement | 1

5. Secondary Outcome: Mucosal Anatomic Recovery
Description: as for outcome 3
Time Frame: 5 weeks after starting treatment with the study product
Population: Only 1 patient had endoscopic evaluation during this time window.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 1
Participants
  Partial improvement | 1
  Complete response | 0

6. Secondary Outcome: Mucosal Anatomic Recovery
Description: as for outcome 3
Time Frame: 6 to 7 weeks after starting treatment with the study product
Population: Only 3 patients had endoscopic evaluation during this time window.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 3
Participants
  Partial improvement | 0
  Complete response | 3

7. Secondary Outcome: Mucosal Anatomic Recovery
Description: as for outcome 3
Time Frame: 9 to 11 weeks after starting treatment with the study product
Population: Only 4 patients had endoscopic evaluation during this time window.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 4
Participants
  Partial improvement | 2
  Complete response | 2

8. Secondary Outcome: Recurrent or Progressive Malignancy
Description: Recurrence or progression of the malignant disease that was the reason for hematopoietic cell transplantation
Time Frame: 2 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants | 1

9. Secondary Outcome: Non-relapse Mortality
Description: Death without prior recurrent or progressive malignancy after transplantation.
Time Frame: 2 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants | 13

10. Secondary Outcome: Survival
Description: Patients who were alive at the specified time after enrollment
Time Frame: 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants | 10

11. Secondary Outcome: Survival
Description: Patients who were alive at the specified time point
Time Frame: 1 year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants | 8

12. Secondary Outcome: Survival
Description: Patients who were alive at the specified time point
Time Frame: 2 years after enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Arm I: Patients received oral lithium carbonate once or twice daily. Treatment continued for up to 8 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I
Number analyzed (Participants) | 20
Participants | 7

13. Secondary Outcome: Causes of Death
Description: Medical condition that made the greatest contribution in causing death
Time Frame: up to 6 years after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants
  Recurrent or progressive malignancy | 2
  Acute graft-versus-host disease | 11
  Chronic GVHD with bronchiolitis obliterans | 2
  Infection | 7
  Multiorgan failure | 2
  Diffuse alveolar hemorrhage | 1
  Hemolytic uremic syndrome | 1

14. Other Pre Specified Outcome: Agents Added to Treat GVHD More Than 3 Days After Enrollment
Description: Any systemic medication given in an effort to control graft-versus-host disease
Time Frame: Up to 100 days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Patients
Number analyzed (Participants) | 20
Participants
  Methotrexate | 1
  Pentostatin | 1
  Rabbit anti-thymocyte globulin | 5
  Mycophenolate mofetil | 4
  Tacrolimus | 2
  Infliximab | 4
  Etanercept | 1
  Alemtuzumab | 1
  Sirolimus | 6

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Treated Patients
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Patients (N=20)
Graft-versus-host disease (Immune system disorders) | 7
Infection (Infections and infestations) | 7
Altered mental status (Nervous system disorders) | 2
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Recurrent malignancy (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated Patients (N=20)
Somnolence or fatigue (Nervous system disorders) | 6
Confusion (Nervous system disorders) | 3
Polyuria (Renal and urinary disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Nausea or vomiting (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
This trial was not controlled in any scientifically valid sense of the term. Clinical management included many changes of treatment other than the use of the study product. The trial had no validated external benchmark for comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No